CLINICAL TRIAL: NCT03122405
Title: Performance Equivalence of Rainbow Acoustic Monitoring (RAM) Small Sensor and RAM Revision D Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR29836A-TP16846C
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test group (Experimental): The subjects will be enrolled in the test group and will simultaneously receive both RAM sensors.
  Interventions: Device: RAM sensors

INTERVENTIONS:
Device: RAM sensors — Noninvasive acoustic monitoring device

SUMMARY:
The purpose of this study was to conduct a side by side comparison of the accuracy of respiratory rate (RR) between our investigational Rainbow Acoustic Monitoring (RAM) small sensor and the FDA-cleared RAM Revision D sensor in healthy volunteers under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Physical status of ASA I or II
* Must be able to read and communicate in English
* Has signed written informed consent

Exclusion Criteria:

* ASA physical status of III, IV, and V
* Subject has any medical condition which in the judgement of the investigator, renders them inappropriate for participating in this study
* Inability to tolerate sitting still or minimal movement for at least 30 minutes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2015-10-29 (Actual); Study Completion 2015-10-29 (Actual)

PRIMARY OUTCOMES:
Performance comparison of RAM sensors by ARMS calculation | 50 minutes
  Performance comparison was determined by comparing the noninvasive respiration rate measurement of the RAM sensors and calculating the arithmetic root mean square (Arms) error value.

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States